CLINICAL TRIAL: NCT04339751
Title: The Effect of Vorinostat on ACTH Producing Pituitary Adenomas in Cushing's Disease
Brief Title: Effect of Vorinostat on ACTH Producing Pituitary Adenomas in Cushing s Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200019; 20-N-0019
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cushing's Disease
Keywords: SAHA; CD
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Vorinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single center, prospective pilot study (Experimental): effectiveness of vorinostat to reduce midnight ACTH levels in patients with Cushing s Disease
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Administration of Vorinostat

SUMMARY:
Background:

Cushing s disease is caused by excess ACTH hormone release by a benign tumor of the pituitary gland. It can lead to decreased quality of life and early death. The current best treatment for Cushing s disease is surgery. If surgery does not work or if the tumor returns, there are no more good treatment options. Vorinostat, which is approved to treat a type of lymphoma, might be a treatment option.

Objective:

To test vorinostat to see if it can kill tumor cells and change the number of hormones released in people with Cushing s disease.

Eligibility:

People ages 18 and older who have Cushing s disease and are scheduled for surgery under protocol 03-N-0164 to remove a tumor in their pituitary gland

Design:

Participants will be screened under protocol 03-N-0164.

Participants will stay in the hospital for 8 days before their surgery.

On the first day, participants will have a physical exam and blood tests. They will have their urine collected for testing all day. They will have an ECG: For this, small metal disks or sticky electrode pads will be placed on their chest to record heart activity.

For the next 7 days, participants will have blood tests and all-day urine collection. They will drink at least 2 liters of fluid per day. They will take the study drug by mouth each morning.

On the eighth day, participants will have their surgery. Leftover tissue will be collected for research.

On the day they are discharged from the hospital, participants will have a physical exam and blood tests.

DETAILED DESCRIPTION:
Study Description

This is a single center, prospective pilot study of effectiveness of vorinostat to reduce midnight ACTH levels in patients with Cushing s Disease. Surgery for resection of ACTH producing pituitary adenoma will be offered at the NIH under another protocol (03-N-0164) as part of standard clinical care. Eligible subjects will be admitted to the Clinical Center for one week prior to surgery, during which time oral vorinostat will be administered daily.

Objectives

Cushing s disease is caused by excess ACTH hormone release by a benign tumor of the pituitary gland. The resulting increase in cortisol levels caused by increased ACTH causes a severe condition that leads to decreased quality of life and early death. The current best first treatment for Cushing s disease is surgery. However, if surgery is unsuccessful or if the tumor returns, there are no good treatment options for patients. In laboratory studies, we discovered that a previously FDA approved oral medication Vorinostat was able to kill tumors cells and reduce ACTH secretion. We want to test whether this drug can be used in patients with Cushing s disease to reduce ACTH levels.

Primary Objective: to determine whether vorinostat reduces midnight plasma ACTH level

Secondary Objectives: to evaluate the effect of vorinostat on urine cortisol levels

Endpoints

Primary Endpoint: midnight plasma ACTH level on the last day of drug administration. Secondary Endpoints: serum cortisol change during drug administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Adult patients (18 years and older)
* Confirmed biochemical diagnosis of Cushing s disease (primary or recurrent) as evidenced by increased 24-hour urine free cortisol (UFC), normal or increased morning plasma Adrenocorticotropic Hormone (ACTH), and pituitary origin of excess ACTH.
* Surgical candidate for resection of ACTH producing pituitary adenoma
* Enrolled in 03-N-0164, Evaluation of Neurosurgical Disorders.
* Able to provide written informed consent at the time of study enrollment.
* Participants who are physically able to become pregnant must use an effective form of birth control from 14 days prior to enrollment through 6 months following the last dose of vorinostat. Participants who are able to father a child must use an effective form of birth control from Day 0 through 3 months following the last dose of vorinostat.

EXCLUSION CRITERIA:

* Patients who have been previously treated with vorinostat.
* Patients who have received sellar radiation.
* Significant medical illnesses that in the investigator s opinion cannot be adequately controlled or would compromise the patient s ability to tolerate this vorinostat.
* Any history of cancer, unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
* History of thromboembolic disorder or deep vein thrombosis
* Presence of abnormal hematological and biochemical parameters, (such as anemia or thrombocytopenia) as defined as:

  * Neutrophil count < 1.5 K//micro L
  * Hemoglobin < 8.0 g/dL.
  * Hematocrit < 0.75x LLN (lower limit of normal)
  * RBC count < 0.75x LLN
  * Platelet count < 100 x 10^3 cells/micro L.
  * Prothrombin time-international normalized ratio (PT-INR) > 1.5x ULN or Activated partial thromboplastin time (aPTT) > 1.5x ULN, with the exception of patients on prophylactic anticoagulation therapy
  * Serum bilirubin level > 1.5x ULN.
* Active infection being currently treated with systemic antibiotics.
* Serious concurrent medical illness including renal failure (creatinine >3.0x - 6.0x ULN) liver failure (ALT/AST >5.0x - 20.0x ULN) or severe cardio-respiratory disease.
* Pregnancy or lactation.
* Presence of any disease that will obscure toxicity or dangerously alter drug metabolism (such as uncontrolled diabetes or bleeding disorders)
* Currently receiving other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat, such as valproate.
* Currently taking another HDACi, such as valproate.
* Currently taking coumadin or its derivative anticoagulants.
* Currently taking any other medication to reduce cortisol or ACTH levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Midnight Plasma ACTH | Day -1, Day 0-1, Day 2, Day 4-6, Discharge
  Relative change in midnight plasma ACTH. Dichotomized relative change using 20% as a cutoff (which is considered as clinical important): relative change >20% for reduction and relative change <=20% for no change).

SECONDARY OUTCOMES:
Urinary Free Cortisol | Day -1, Day 0-1, Day 2, Day 4-6, Discharge
  Relative change in 24-hour urinary free cortisol during 7 day administration of Vorinostat

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Chittiboina, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. we will share all IPD that results in a publication on a public repository, as required by most journals. the data will be de-identified and anonymized.

REFERENCES:
- [Background] Arnaldi G, Angeli A, Atkinson AB, Bertagna X, Cavagnini F, Chrousos GP, Fava GA, Findling JW, Gaillard RC, Grossman AB, Kola B, Lacroix A, Mancini T, Mantero F, Newell-Price J, Nieman LK, Sonino N, Vance ML, Giustina A, Boscaro M. Diagnosis and complications of Cushing's syndrome: a consensus statement. J Clin Endocrinol Metab. 2003 Dec;88(12):5593-602. doi: 10.1210/jc.2003-030871. PMID 14671138
- [Background] Cushing H. The basophil adenomas of the pituitary body and their clinical manifestations (pituitary basophilism). 1932. Obes Res. 1994 Sep;2(5):486-508. doi: 10.1002/j.1550-8528.1994.tb00097.x. No abstract available. PMID 16353601
- [Background] Newell-Price J, Bertagna X, Grossman AB, Nieman LK. Cushing's syndrome. Lancet. 2006 May 13;367(9522):1605-17. doi: 10.1016/S0140-6736(06)68699-6. PMID 16698415
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-N-0019.html